CLINICAL TRIAL: NCT05460429
Title: An Open Clinical Trial to Evaluate Immunogenicity,Safety and Protective Effect of Live Attenuated Varicella Vaccine and a Clinical Trial on Antibody Level and Etiology of Varicella Zoster Virus in Zhejiang Province
Brief Title: Immunogenicity, Safety and Protective Effect of Live Attenuated Varicella Vaccine and Study on Antibody Level and Etiology of Varicella Zoster Virus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VAR-MA4002-ZJ
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-04

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Immunogenicity and safety group (Experimental): 360 subjects including 120 subjects aged 1-3 years with no history of varicella vaccination,240 subjects aged 4-6 years with a history of 1 dose of varicella vaccine will be enrolled to evaluate the immunogenicity and safety of varicella vaccine.All subjects will receive one dose of varicella vaccine.
  Interventions: Biological: Live attenuated varicella vaccine
- Antibody level investigation study group (Experimental): Immunization levels will be monitored among 2530 subjects aged 0-59 years old and will be collected venous blood to detect varicella antibody.
  Interventions: Biological: Live attenuated varicella vaccine
- Safety group (Experimental): 30000 subjects aged 1-12 years old will be enrolled to conduct safety observation of mass vaccination of varicella vaccine.All subjects will receive one dose of varicella vaccine and all adverse events of all subjects will be collected.
  Interventions: Biological: Live attenuated varicella vaccine
- Protective effect group (Experimental): 5000 subjects aged 1-12 years old will be enrolled to conduct protective effect study of varicella vaccine after exposure.
  Interventions: Biological: Live attenuated varicella vaccine
- Etiology Group (Experimental): 30 varicella cases aged 1-12 years old from study 4 will be enrolled. Herpes fluid or pharyngeal swab samples of subjects will be collected to study the pathogenicity of varicella.
  Interventions: Biological: Live attenuated varicella vaccine

INTERVENTIONS:
Biological: Live attenuated varicella vaccine — The live attenuated varicella vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. Live attenuated varicella-virus in 0.5 mL injection water with sucrose,sodium glutamate,sodium chloride,potassium chloride, sodium dihydrogen phosphate, potassium dihydrogen phosphate per injection.The routine of administration is intramuscular injection into deltoid region of the lateral upper arm. And the immunization schedule is one dose of live attenuated varicella vaccine on day 0.

SUMMARY:
This is Phase 4 clinical trial of live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd .The purpose of this study is to evaluate the immunogenicity and safety of a single dose of varicella vaccine in healthy children aged 1-6 years with different varicella immunization histories, to evaluate the antibody level of varicella-zoster virus in healthy people aged 0-59 years in Zhejiang Province.

DETAILED DESCRIPTION:
This study is Phase Ⅳ clinical trial.The experimental vaccine manufactured by Sinovac(Dalian) Vaccine Technology Co., Ltd.This clinical trial consists of five parts,and A total of 37920 subjects will be enrolled.

Study 1,360 subjects including 120 subjects aged 1-3 years with no history of varicella vaccination ,240 subjects aged 4-6 years with a history of 1 dose of varicella vaccine will be enrolled to evaluate the immunogenicity and safety of varicella vaccine.All subjects will receive one dose of varicella vaccine.

Study 2,2530 subjects aged 0-59 years old will be enrolled and will be collected venous blood to detect varicella antibody and conduct investigation of varicella antibody level in healthy people.

Study 3,30000 subjects aged 1-12 years old will be enrolled to conduct safety observation study.All subjects will receive one dose of varicella vaccine and all adverse events of all subjects will be collected.

Study 4,5000 subjects aged 1-12 years old will be enrolled to conduct protective effect study of varicella vaccine after exposure.

Study 5,30 subjects aged 1-12 years old will be enrolled. Herpes fluid or pharyngeal swab samples of subjects will be collected to study the pathogenicity of varicella.

ELIGIBILITY:
Unified Inclusion Criteria:

* Participants aged 1-12 years ;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8-12 years, both subjects and guardians need to sign the informed consent form) and be able to follow all research procedures;
* Proven legal identity.

Special Inclusion Criteria for each study:

Inclusion criteria of the study population for immunogenicity and safety evaluation of varicella vaccine:

* Be able to participate in the whole process of vaccination and blood collection;
* Healthy children aged 1-3 years with no history of varicella vaccination;
* Healthy children aged 4-6 years with a history of 1 dose of varicella vaccine.

Inclusion criteria for investigation of varicella antibody level:

* Healthy people aged 0-59 years and participate voluntarily for the study;
* Have no serious chronic disease or acute disease;

Inclusion criteria of the study population for safety evaluation of varicella vaccine mass vaccination:

* Participants aged 1-3 years with no history of varicella vaccination;
* Participants aged 4-12 years with no history of varicella vaccination or with a history of 1 dose of varicella vaccine.

Inclusion criteria of study population for protective effect of varicella vaccine after exposure:

* Children aged 1-12 years exposed to varicella outbreaks;
* History with no varicella or shingles;

Inclusion criteria of study population for etiological study on the pathogenic strains of varicella cases:

* Clinical cases of varicella consent for herpes zoster or pharyngeal swab collection.

Exclusion Criteria:

* History of 2 doses of varicella vaccination;
* Previous history of varicella or herpes zoster (not applicable to investigation of varicella antibody level);
* History of severe allergic reactions to vaccines (e.g.acute anaphylaxis, angioneurotic edema, dyspnea, etc.);
* Suffering from acute disease or acute episode of chronic disease;
* Any confirmed or suspected immunodeficiency disease, including human immunodeficiency virus (HIV) infection;
* Axillary temperature >37.0°C;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 28 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Max Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37920 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
GMT of varicella antibody in children aged 1-6 years | 30 days after vaccination
  GMT of varicella antibody at 30 days after vaccination of varicella vaccine in children aged 1-6 years.
GMT of varicella antibody in healthy people aged 0-59 years | 30 days after vaccination
  GMT of varicella antibody at 30 days after vaccination in different age groups of healthy people aged 0-59 years.

SECONDARY OUTCOMES:
Seroconversion rates of varicella antibody in children aged 1-6 years | 30 days after vaccination
  Seroconversion rates of varicella antibody at 30 days after vaccination of varicella vaccine in children aged 1-6 years.
GMI of varicella antibody in children aged 1-6 years | 30 days after vaccination
  GMI of varicella antibody at 30 days after vaccination of varicella vaccine in children aged 1-6 years.
Incidence of adverse reactions at 24 hours after vaccination | 24 hours after vaccination
  Incidence of adverse reactions at 24 hours after vaccination of varicella vaccine in children aged 1-6 years
Incidence of adverse reactions at 3 days after vaccination | 3 days after vaccination
  Incidence of adverse reactions at 3 days after vaccination of varicella vaccine in children aged 1-6 years
Incidence of adverse reactions at 14 days after vaccination | 14 days after vaccination
  Incidence of adverse reactions at 14 days after vaccination of varicella vaccine in children aged 1-6 years.
Incidence of adverse reactions at 30 days after vaccination | 30 days after vaccination
  Incidence of adverse reactions at 30 days after vaccination of varicella vaccine in children aged 1-6 years.
Incidence of adverse reactions at 14 days after mass vaccination | 14 days after mass vaccination
  Incidence of adverse reactions at 14 days after mass vaccination of varicella vaccine in children aged 1-12 years
Incidence of adverse reactions at 30 days after mass vaccination | 30 days after mass vaccination
  Incidence of adverse reactions at 30 days after mass vaccination of varicella vaccine in children aged 1-12 years
seropositive rates of varicella antibody | 30 days after vaccination
  Seropositive rates of varicella antibody at 30 days after vaccination in all age groups of healthy people.

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Zhejiang Provincial Center for Disease Prevention and Control
Locations (3):
- China (3):
  - Laian Center for Disease Control and Prevention, Chuzhou, Anhui
  - Liandu District Center for Disease Control and Prevention, Lishui, Zhejiang
  - Jiangshan Center for Disease Control and Prevention, Quzhou, Zhejiang